CLINICAL TRIAL: NCT05966207
Title: Making a Difference 3 - Individual Intervention of Cognitive Stimulation
Brief Title: Individual Intervention of Cognitive Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Escola Superior de Enfermagem de Coimbra (Other)
Responsible Party: Principal Investigator, Joao Apostolo, PhD, Escola Superior de Enfermagem de Coimbra
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: FD3-2022
Record Dates: First submitted 2023-07-21; First posted 2023-07-28 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Cognitive Dysfunction
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Individual Cognitive Stimulation (Experimental): The Individual Cognitive Stimulation (ICS) program to be implemented is called "Making a Difference 3 - Individual Intervention of Cognitive Stimulation - A manual for caregivers" (MD3). It was specifically designed to be applied in a home context, with informal/family caregivers taking charge of implementing the stimulation sessions (Apostolo, Silva, Costa & Bobrowicz-Campos, 2019; Yates et al., 2015). The MD3 program has been translated and validated for the Portuguese culture and language (Silva, 2019).
  Interventions: Behavioral: Individual Cognitive Stimulation

INTERVENTIONS:
Behavioral: Individual Cognitive Stimulation — The Individual Cognitive Stimulation will be conducted by caregivers, with support by the research team. The intervention will span 12 weeks, consisting of three weekly sessions (30 minutes each session), totaling 36 sessions. Caregivers in this study will utilize a previously translated and validated version of "Making a Difference 3 - Individual Intervention of Cognitive Stimulation - A manual for caregivers," specifically adapted for the European Portuguese population.

SUMMARY:
Population aging in Portugal has led to problematic social issues (American Psychiatric Association, 2013; Spector, Woods & Orrell, 2008; Wimo & Prince, 2010). At the same time, there is a noticeable increase in the prevalence of Neurocognitive Disorders (NCDs), commonly referred to in clinical practice as mild cognitive impairment and dementia (Apóstolo, Cardoso, Silva & Costa, 2014; Apóstolo & Cardoso, 2014).

NCDs can be classified based on the degree of cognitive decline, ranging from mild to major, and based on etiology, which includes Alzheimer's disease, Vascular dementia, Lewy body dementia, Frontotemporal dementia, and others (American Psychiatric Association, 2013).

In the European context, Portugal is among the minority of countries that do not have an official strategy for the care of people with mild cognitive impairment and dementia. Therefore, it is imperative to define national health policies that address the identified needs (Knapp et al., 2006).

Currently, non-pharmacological interventions, such as Individual Cognitive Stimulation (ICS), are gaining relevance as treatment responses to the aforementioned syndromes, due to the increasing clinical, social, and economic impact of mild cognitive impairment and dementia (Aguirre, Hoare, Spector, Woods, & Orrell, 2014; Apóstolo et al., 2014).

ICS can be considered the implementation of a set of meaningful activities, carried out over several sessions, usually in a social context, with the aim of stimulating various domains, including attention, thinking, language, memory, and calculation (Aguirre et al., 2012; Apóstolo et al., 2014; Yates, Orrell, Spector & Orgeta, 2015).

Current evidence supports the effectiveness of this intervention, indicating that ICS programs are associated with health benefits, particularly in cognition, mood, well-being, functional activity, quality of life, and communication skills (Apóstolo et al., 2014; Yates et al., 2014).

Providing care to people with mild cognitive impairment and dementia poses a challenge for the healthcare system, necessitating the implementation of specific interventions to increase self-care potential, autonomy, adaptation, and coping with deficits, as well as empowering the family and/or support network (Alzheimer Europe, 2013; Orrell et al., 2012; Woods, Aguirre, Spector & Orrell, 2012; Yates et al., 2015). Due to the global pandemic context of SARS-CoV-2, social care institutions for the elderly underwent changes in their dynamics. One of the measures implemented during the emergency plan was the closure of adult day care centers. The elderly who previously attended these social care facilities are now staying in their own homes or with family/informal caregivers, thus being deprived of the social and cognitive stimuli they were accustomed to.

The mobilization of this population to their homes has led to increased social isolation and loneliness, which are underestimated public health risks. These factors affect a significant proportion of the elderly population and can lead to cognitive decline, feelings of loneliness, sadness, and abandonment, which were previously alleviated by the social care centers (National Academies of Sciences, Engineering, and Medicine, 2020).

Given the described situation, the Making a Difference 3 program - an ICS program - represents an excellent implementation option, as it can be developed in various contexts, including the home environment, using cost-effective resources, addressing many of the needs of both individuals with cognitive impairment and their informal family caregivers.

In summary, in Portugal, there is no established practice of implementing structured ICS interventions with individual sessions for use in the home environment. Thus, there is a need for the MD3 program to be disseminated to promote best practices. In response to the needs arising from the current pandemic context, the team of this project aims to produce national evidence on the effect of ICS in individuals with mild cognitive impairment and dementia, in the home environment of the elderly person, managed by informal caregivers and supervised by healthcare professionals.

ELIGIBILITY:
Inclusion Criteria:

* Older adults or near-elderly individuals (aged 60 years or above), diagnosed with mild cognitive impairment or dementia by a neurology or psychiatry specialist, or validated by a family physician based on DMS-III/IV/5 or ICD-9/10 criteria;
* Without significant physical illness or disability.
* Having an informal caregiver, whether a family member, friend, neighbor, or volunteer.
* Presence of mild to moderate cognitive impairment according to the 6-Item Cognitive Impairment Test (6CIT), translated and adapted by Apóstolo and Paiva (2015).
* Individuals with mild cognitive impairment or dementia who are capable of communication and understanding.
* Individuals residing in the community (at home).
* Having an available informal caregiver, whether a family member, friend, neighbor, or volunteer, who is capable of implementing the individual cognitive stimulation program.

Exclusion Criteria:

* Elderly individuals or informal caregivers with a history of serious psychiatric illness diagnosed before the age of 60 are excluded from participation.
* Informal caregivers with any level of cognitive impairment, even mild (according to DSM-5 criteria), are not eligible for inclusion.
* Elderly individuals residing in a social response facility, such as a nursing home or elderly residence, are not considered for this study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2021-12-27 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Cognition | Assessed at baseline (week 0, pre-intervention) and week 13 (post-intervention)
  Assessed using the Saint Louis University Mental Status Test (SLUMS), by Tarik et al. (2006)
Quality of Life | Assessed at baseline (week 0, pre-intervention) and week 13 (post-intervention)
  Assessed using the Quality of Life in Alzheimer's disease (QoL-AD) scale by Logsdon et al. (1999)

SECONDARY OUTCOMES:
Dementia-related behavioral symptoms | Assessed at baseline (week 0, pre-intervention) and week 13 (post-intervention)
  Assessed using The Neuropsychiatric Inventory (NPI) by Cummings et al. (1994)
Quality of the Carer-Patient Relantionship | Assessed at baseline (week 0, pre-intervention) and week 13 (post-intervention)
  Assessed using the Quality of the Carer-Patient Relationship (QCPR) scale by Spruytte et al. (2002), validated to the European Portuguese population by Silva et al. (2019)

CONTACTS AND LOCATIONS:
Locations (1):
- The Health Sciences Research Unit: Nursing, Coimbra, Portugal

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data (IPD) will be made available upon reasonable request made to the principal investigator.